CLINICAL TRIAL: NCT06102122
Title: To Evaluate the Acceptability (including Gastrointestinal Tolerance and Compliance) of an Adult Tube-feed Formula with Ingredients Derived from Food.
Brief Title: Acceptability and Tolerance Study of Adult Tube Feed with Food with Food Derived Ingredients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Compleat 001
Record Dates: First submitted 2023-08-22; First posted 2023-10-26 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-04

CONDITIONS: Dietary Exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients well established on tube feeds will act as their own control (Other): Patients will switch from current to new tube feed.
  Interventions: Dietary Supplement: Compleat

INTERVENTIONS:
Dietary Supplement: Compleat — Patients well established and stable on a standard enteral tube feed with food derived ingredients will act as their own controls and make a product switch

SUMMARY:
Product acceptability data from 15 participants are required in order to submit an application to the Advisory Committee on Borderline Substances (ACBS) and the Health Service Executive (HSE) submission for Ireland for product registration.

DETAILED DESCRIPTION:
To evaluate the acceptability (including gastrointestinal tolerance and compliance) of an adult tube-feed formula with ingredients derived from food for the dietary management of participants who require a tube feed. .

The acceptability data from 15 participants will be collected in order to submit an application to the Advisory Committee on Borderline Substances (ACBS) and the Health Service

Executive (HSE) for Ireland. Participants will be provided with one month supply of tube feed and will be asked to complete a daily diary and short questionnaire to record information allowing assessment of the following:

* Gastrointestinal tolerance
* Compliance with prescribed feed volumes

ELIGIBILITY:
Inclusion Criteria:

* Require a tube feed (taking >75% of energy needs from their feeding tube) as part of their dietary management for disease related malnutrition
* Adults and children requiring an adult enteral formula as assessed by the dietitian.
* Patients well-established and stable on a standard formula or currently on Isosource® Junior Mix.
* Willingly given, written, informed consent from patient or consultee. For those who lack capacity to provide formal consent for themselves, this may be provided by a personal or consultee in accordance with the Mental Capacity Act.
* Willingly given, written assent (if appropriate) on behalf of patients under 18.

Exclusion Criteria:

* Inability to comply with the study protocol, in the opinion of the investigator
* Known food allergies to any ingredients (see ingredients list)
* Patients with significant renal or hepatic impairment - Change in current medication or use of additional macro/micronutrient supplements during the study period, unless clinically indicated and prescribed by the investigator (must be recorded in patient case record file).
* Participation in another interventional study within 2 weeks of this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Daily record via participant diary | 7 days
  Daily Gastrointestinal diary as questionnaire, increase, decrease or no change
Formula intake diary | 28 days
  mL per day

CONTACTS AND LOCATIONS:
Overall Officials: Tanita Flood, Principal Investigator — Royal Hospital for Neuro-disability; Martha Van der Linde, Principal Investigator — Community Paediatric Dietitian Worcestershire, Hastings UK; Minal Patel, Principal Investigator — Barts and London Hospital Trust London UK; Adrian Gilson, Principal Investigator — Newham General Hospital London UK
Locations (1):
- Tanita Flood, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Will upload the data as it becomes available